CLINICAL TRIAL: NCT01722084
Title: Community-embedded Reproductive Health Care for Adolescents in Latin America (CERCA).
Brief Title: Community-embedded Reproductive Health Care for Adolescents in Latin America.
Acronym: CERCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Lithuanian University of Health Sciences (Other); VU University of Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011/380; FP7-health-241615
Record Dates: First submitted 2012-10-29; First posted 2012-11-06 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Sexual and Reproductive Health Problems
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community-eùbedded reproductive health interventions (Experimental): Members of communities that belonged to the intervention arm were exposed to complex interventions addressing different target groups (adolescents, parents, authorities and health providers) and focusing on various behaviours that were related to communication about sexuality, information seeking, access to health care and safe sexual intercourse.
  Interventions: Behavioral: Theory of planned behaviour (TPB) and social cognitive theory (SCT).
- Community members without intervention (No Intervention)

INTERVENTIONS:
Behavioral: Theory of planned behaviour (TPB) and social cognitive theory (SCT). — TPB is appropriate to influence adolescents' behaviour related to the use of contraceptive methods and their health/information seeking behaviour. The SCT helped to find out strategies to improve communication about sexuality, to promote openness towards adolescents' sexuality among parents, community members and health providers and for health providers to adopt a more adolescent friendly attitude.The development of the strategies in the different countries is a dynamic process that is continuously being adapted. The target groups were "driving" the process of identifying, selecting and implementing interventions. Therefore, local institutions were involved in the intervention. Attention was paid to ensure that the interventions were in line with the existing local structures/policies and reinforce the local health system.Primary health care services had a key role in the interventions. Gender was a transversal topic throughout the intervention process.
  Arms: Community-eùbedded reproductive health interventions

SUMMARY:
Adolescents in Latin America are at major risk for unwanted pregnancies leading to unsafe abortions and maternal health risks. Mostly, adolescent health programmes tend to focus on unidirectional interventions aiming at a single determinant of adolescents´ sexual and reproductive health. However, evidence exists that a complex health problem should be addressed by an equally nuanced and multipronged response. Knowledge is lacking on how to develop a comprehensive approach to promote adolescents' sexual health.

The CERCA study will conduct an implementation based on the hypothesis that a comprehensive strategy of community-embedded interventions helps to improve the sexual health of adolescents. We will test this hypothesis and describe the development, implementation and testing of interventions in three Latin American cities: Cochabamba (Bolivia), Cuenca (Ecuador) and Managua (Nicaragua).

The research methodology has been designed based on the methodological frameworks of action research, community based participatory research and intervention mapping.

The interventions are complex addressing different target groups (adolescents, parents, authorities and health providers) and focussing on various behaviours that are related to communication about sexuality, information seeking, access to health care and safe sexual intercourse.

For the evaluation of effectiveness a randomised and non-randomised controlled study was developed for respectively Managua and the two other cities. Furthermore a process evaluation is conducted.

This research will result in a framework that will contribute to the planning of interventions that are effective and responsive to adolescents' sexual health needs.

ELIGIBILITY:
Inclusion Criteria:

Nicaragua - adolescents aged 13-18 living in the 33 town districts of Managua with a population number that varies between 1400 and 4500 inhabitants and with more than 50 % poor people.

Bolivia and Ecuador: Students from conveniently selected secondary schools in Cochabamba (Bolivia) and Cuenca (Ecuador).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9625 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Self-reported use of modern contraceptives at 18 months of interventions. | At 18 months of intervention
  Self-reported exposure to intervention activities and registered participation at intervention activities.

SECONDARY OUTCOMES:
Self-reported ease to communicate about sexuality with parents, partner, friends. | At 18 months of intervention
  Self-reported exposure to intervention activities, registered participation at intervention activities and registered access of adolescents to health services.
Self-reported access health services for sexual and reproductive health. | At 18 months of intervention
  Self-reported exposure to intervention activities, registered participation at intervention activities and registered access of adolescents to health services.
Self-reported information seeking behaviour. | At 18 months of intervention
  Self-reported exposure to intervention activities, registered participation at intervention activities and registered access of adolescents to health services.
Self-reported pregnancy. | At 18 months of intervention
  Self-reported exposure to intervention activities, registered participation at intervention activities and registered access of adolescents to health services.

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Temmerman, MD, PhD, Principal Investigator — University Ghent
Locations (4):
- South Group, Cochabamba, Bolivia
- Universidad de Cuenca, Cuenca, Ecuador
- Nicaragua (2):
  - Centro de investigaciones y estudios de salud, Managua
  - Instituto Centro Americano de la Salud, Managua

REFERENCES:
- [Derived] Decat P, Nelson E, De Meyer S, Jaruseviciene L, Orozco M, Segura Z, Gorter A, Vega B, Cordova K, Maes L, Temmerman M, Leye E, Degomme O. Community embedded reproductive health interventions for adolescents in Latin America: development and evaluation of a complex multi-centre intervention. BMC Public Health. 2013 Jan 14;13:31. doi: 10.1186/1471-2458-13-31. PMID 23311647